CLINICAL TRIAL: NCT00156689
Title: A Pilot Study in a Double Blind, Randomized, Placebo-Controlled, Parallel-Group, 16 Week, Trial Design Evaluating the Efficacy and Safety of Levetiracetam 500 mg Tablets in Bid Administration (Daily Dose Ranging From 1000 mg to 3000 mg), in Adults (>18 Years of Ages) Suffering From Chronic Idiopathic Axonal Polyneuropathy
Brief Title: A Study to Determine if Levetiracetam Will Assist Those Suffering From Chronic Idiopathic Axonal Polyneuropathy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Gary Duncan, M.D., Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050465; NCT00298948 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Idiopathic Axonal Polyneuropathy
Keywords: polyneuropathy
MeSH Terms: conditions — Polyneuropathies | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levetiracetam

SUMMARY:
Considering the mechanisms of action which provide efficacy in epilepsy, it is hypothesized that treatment with levetiracetam will reduce the neuronal excitability involved in neuropathic pain associated with CIAP. Thus, there is a potential for levetiracetam to bring therapeutic benefit for the subjects because of its specific mechanism of action, its safety profile and the absence of interaction with other drugs.

DETAILED DESCRIPTION:
Based on literature and expert opinion, and despite the efforts made to better treat the spectrum of neuropathic pains, there are still unmet needs. The available treatments are not effective as monotherapy administration in the vast majority of patients and polypharmacy with several medications is often necessary. Tricyclic antidepressants (TCAs), mainly amitriptyline, are still a mainstay of treatment for painful peripheral neuropathy, but at the risk of some dose-limiting adverse events, which may reduce their effectiveness. TCA treatment effect is inconsistent and limited by side effects. In one clinical trial while about 50% of patients achieved significant or complete relief of pain 81% experienced side effects and in 71% the side effects were dose limiting. TCAs can produce sedation, urinary retention, and orthostatic hypotension that are of particular concern in the elderly and patients with cardiovascular disease. In the same study desipramine was associated with a slightly lower rate of side effects it offered only 40% of patients significant or complete relief of neuropathic pain. Fluoxetine was no more effective than placebo in pain relief. (Max, 1992). Due to the scarcity of controlled clinical trials and the inconclusive results of available trials, physicians vary markedly in their suggested regimens for neuropathic pain management. (Beydoun, 1999).

Antiepileptic drugs are being used more frequently in non-epileptic indications such as neuropathic pain. One of the mechanisms by which neuropathic pain occurs is related to an increased excitability of central neurons. Although their precise mechanism of action in neuropathic pain remains unknown, antiepileptic drugs are believed to exert their antineuralgic activity by suppressing the neuronal hyperexcitability state that characterizes neuropathic pain. A small crossover trial of carbamazepine produced clinical benefit is a significant number of patients but with side effects of somnolence in 50%, dizziness in 40% and rash in 6% (Rull, 1969). Gabapentin showed benefit over placebo in a 165-subject randomized study of painful diabetic neuropathy pain; side effects were noted to be mild or moderate in most but 8% withdrew due to side effects (Backonja, 1998). In a placebo controlled study of lamotrigine in diabetic neuropathy there was s significant reduction in daily pain scores compared to placebo; side effects were noted in about half of the treated group but were minor. (Eisenberg, 2001). Results of treatment trials sing valproate in painful diabetic neuropathy have been variable with both positive (Kochar, 2004) and negative trials (Otto, 2004). Treatment of neuropathic pain in chronic idiopathic axonal polyneuropathy has received limited study. In a single open label study or CIDP pain tiagabine produced about 30% reduction in pain severity but almost half of the patients discontinued the trial (Novak, 2001).

Levetiracetam has been tested in two animal models of neuropathic pain (Ardidd, 2001). In the streptozocin diabetic rat model, reactivity to a pressure on the paw was assessed and revealed that the ED50 for levetiracetam was comparable to the one observed in the epilepsy models. Further, hyperalgesia was dose-dependently decreased by levetiracetam. On the other hand, in the mononeuropathic sciatic nerve ligature model, hyperalgesia was not significantly diminished. Carbamazepine is effective in the sciatic nerve ligature model. Animal models of neuropathic pain are considered suggestive of activity in humans but they are not directly predictive.

Based on the data from the animal studies in neuropathic pain models, levetiracetam has been tested in a limited basis in two human types of neurological pain, painful diabetic peripheral neuropathy and sural nerve stimulation in healthy volunteers. The diabetic neuropathy study was a 12-week, multicenter, randomized, placebo-controlled, parallel group study to evaluate the efficacy and safety of flexible dosing with LEV at 500 to 1500 mg bid. A total of 105 subjects were included in the ITT population, 52 subjects in placebo and 53 subjects in the LEV group. At baseline, the treatment groups were comparable with respect to demographic and other baseline characteristics. There were no statistically significant or clinically meaningful treatment differences observed throughout the evaluation period relative to baseline (personal communication).

In the randomized, double-blind, crossover, electrical sural nerve stimulation study, pain was assessed in healthy volunteers before and 2, 4, 6, 8 and 24 hours after 1500 mg levetiracetam or placebo was orally administered. Levetiracetam significantly increased the threshold for pain detection when single electrical sural nerve stimulation was used, but had no effect on temporal pain summation after repetitive sural nerve stimulation (CDC). It has, however, been demonstrated that results from one type of neuropathic pain cannot necessarily be extrapolated to other types, as the negative results of the 1998 study of amitriptyline in HIV-related painful neuropathy demonstrates (Beydoun, 1999).

A small, investigator-initiated open label trial using levetiracetam in postherpetic neuralgia (PHN) was recently completed. The study, published in Neurology, reported 6/10 patients had improvement in PHN symptomatology after a 12-week treatment with levetiracetam. All 10 patients exposed had received multiple prior treatments for PHN (Rowbotham, 2003).

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, the following criteria must be met:

Subject is or has:

* Male or female outpatient greater than or equal to 18 years of age;
* Suffering presently from neuropathic pain, which has been present for at least 3 months and is clinically felt to be associated with CIAP;
* CIAP defined by the following clinical criteria: Primary = distal predominant sensory loss in feet and/or hands; preserved motor strength and deep tendon reflexes; normal routine nerve conduction study velocities and amplitudes; no identifiable etiology after appropriate evaluation; Secondary = neuropathic pain in feet; neuropathic pain in hands; abnormal QSART, age 45-70 years, autonomic dysfunction.
* Neuropathic pain at entry into the study must meet the following criteria: a VAS of at least 40 mm at visit 2 (to assess pain intensity during the past week) and with an average daily score of at least 4 on the PSS during the baseline period as evaluated on a minimum of 4 days;
* An estimated creatinine clearance of at least 80 ml/min. If the subject has a history or symptoms of renal impairment, an estimated creatinine clearance will be obtained at the baseline visit. If the estimated creatinine clearance is </= 80 ml/min the subject is not eligible to participate;
* Capable of understanding and completing diaries and questions, and adhering to the protocol, in the judgment of the investigator;
* Females of childbearing potential must have a negative serum pregnancy test at the selection visit and at Visits 2 - 6 (and a negative result on the accompanying urine pregnancy test at Visit 2). Females must be surgically sterile, postmenopausal for at least 2 years prior to visit 1, must have undergone tubal ligation or using an acceptable method of birth control for the duration of the study (oral contraceptives must be stable for at least one full month prior to visit 1). Abstinence is not an acceptable method of contraception for the study.
* Written informed consent obtained prior to procedures being performed and the consent process documented;
* Able to follow written and verbal instructions in English or in Spanish and be willing to attend the required study visits and complete the required daily assessments (Spanish speaking patients can only be enrolled at sites with staff who are fluent in Spanish);
* A telephone where they can be directly contacted.

Exclusion Criteria:

* Subjects must be excluded if they meet any of the following criteria.

Subject is or has:

* Receiving professional psychological support (such as cognitive behavioral therapy) currently or within 2 weeks prior to visit 1 specifically for coping with PHN;
* Previous neurolytic or neurosurgical therapy for peripheral neuropathy pain, at any time in the subject's history or treatment with TENS (transelectroneuro stimulation) currently or within the past 2 weeks;
* Known co-existent source of pain or painful peripheral neuropathy, (untreated hypoparathyroidism, vitamin B12 deficiency, amyloidosis, connective tissue disease, porphyria, diabetic peripheral neuropathy, complex regional pain syndrome, alcoholism, hepatitis, uremia, syphilis, myeloma, malignancy (less than 5 years in remission), peripheral nerve trauma (including surgery), drug induced peripheral neuropathy (e.g., vinca alkaloids, taxols, etc.) or other systemic disease associated with a secondary painful neuropathy);
* Known significant neurological disorder other than the study disease or a condition which can mimic stroke with distal neurological deficit (amyotrophy, radiculopathy, history of TIAs, multiple sclerosis, or any amputations);
* Conditions known to be associated with immunosuppressive states;
* Significant lactose intolerance;
* Presence of signs or symptoms of rapidly progressing clinically significant brain disorder or dementia;
* Significant and severe medical conditions (such as severe cardiac dysfunction, bone marrow suppression, severe hepatic disease) which may impair reliable participation in the trial;
* Clinically significant deviations from reference range values for laboratory parameters such as hepatic markers (ALAT/SGPT, ASAT/SGOT, alkaline phosphatase, γGT), platelets < 100,000/μl, leukocyte count < 3500/mm3 or neutrophil cells < 1,800/μl;
* Alcohol or drug abuse currently or within the past year according to DSM-IV-TR criteria as interpreted by the investigator;
* Current participation or participation within the last 30 days in another investigational clinical trial or dosing with any non-study drug not approved for use in the United States;
* Clinically significant major depression defined as a Beck Depression Inventory Score > 21 at selection including those with a history of Bipolar Disorder;
* History of suicidal ideation in the past 3 months or suicide attempt within the last 10 years;
* Intake of more than two classes of medications to treat pain at study entry (see Sectio on Concomitant Treatment);
* Intake of levetiracetam within 2 weeks prior to visit 1;
* Currently receiving treatment with a spinal cord stimulator
* Intake of benzodiazepines (for any indication), skeletal muscle relaxants, orally administered steroids, local and topical agents for the relief of peripheral polyneuropathy pain, and anticonvulsant agents within 2 weeks prior to visit 1 or during the study;
* Discontinued treatment with antidepressants < 4 weeks prior to visit 1;
* Current use or use within 2 weeks prior to visit 1 of topical steroids specifically for the treatment of peripheral neuropathy pain;
* Current use or use within 2 weeks prior to visit 1 of lidocaine patches as a therapy for peripheral neuropathy pain, regardless of frequency or duration of use;
* History of hormone replacement therapy which has not been stable and ongoing for at least 2 weeks prior to visit 1;
* A female subject who is currently breast feeding an infant;
* Presence of an indwelling cardiac pacemaker or other indwelling electrical device that would preclude performance of nerve conduction studies.
* Known hypersensitivity to levetiracetam or any of the inactive ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Exploratory efficacy endpoint
The primary exploratory efficacy variable is the absolute change in the average weekly PSS from the baseline period to the last 7 days of the evaluation period (Last Observation Carried Forward).

SECONDARY OUTCOMES:
The secondary exploratory efficacy endpoints and/or analysis methods are:
Reduction of at least 30% in the mean PSS over the last week of the evaluation period compared to the baseline period (30% Responder).
Reduction of at least 50% in the mean PSS over the last week of the evaluation period compared to the baseline period (50% Responder).
Percent change in the mean PSS from the baseline week to each weekly mean.
Absolute change from the baseline week to each weekly mean in the PSS.
Changes from the baseline week to each weekly mean, and to the last week of evaluation period, in the SIS.
Absolute changes from the randomization visit to each evaluation period/early discontinuation visit, in each score (Total pain score, Sensory score, Affective score, Present Pain Intensity (PPI) and VAS) of the SF-MPQ.
Subject Global Impression of Change (SGIC) at visit 6 or the last visit of the evaluation period.
Clinician's Global Impression of Change (CGIC) at visit 6 or the last visit of the evaluation period.

CONTACTS AND LOCATIONS:
Overall Officials: Gary W. Duncan, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States